CLINICAL TRIAL: NCT00008216
Title: The Use Of Peripheral Blood Stem Cells For Allogeneic Transplantation
Brief Title: Blood Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Savage, Professor of Medicine, Columbia University
Other Study IDs: AAAA5571; CPMC-IRB-AAAA5571; CPMC-CAMP-016; NCI-G00-1891
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Adult Langerhans Cell Histiocytosis; Childhood Langerhans Cell Histiocytosis; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; childhood Langerhans cell histiocytosis; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; chronic myelogenous leukemia, BCR-ABL1 positive; Philadelphia chromosome negative chronic myelogenous leukemia; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; intraocular lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; juvenile myelomonocytic leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; chronic myelomonocytic leukemia; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes; adult Langerhans cell histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples Without DNA — Standard bloodwork that would be required for transplantation patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- alloSCT group: Patients undergoing allogeneic blood or marrow stem cell transplantation (alloSCT).
  Interventions: Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: Peripheral Blood Stem Cell Transplantation

SUMMARY:
RATIONALE: Giving chemotherapy drugs and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying the effectiveness of donor peripheral blood stem cell transplant in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and safety of allogeneic peripheral blood stem cell transplantation in achieving engraftment in patients with hematologic malignancy.
* Determine the hematopoietic recovery, incidence of chemoradiotherapeutic toxicity, relapse, graft-versus-host disease, and survival of patients treated with this regimen.

OUTLINE: Patients receive a preparative chemoradiotherapeutic regimen and graft-versus-host disease prophylaxis prior to transplantation. Patients undergo allogeneic peripheral blood stem cell transplantation on day 0.

Patients are followed every 1-2 weeks for 6 months and at 9, 12, 24, and 36 months.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Chronic myelogenous leukemia

    * Philadelphia chromosome-positive OR
    * Molecular evidence of bcr/abl gene rearrangement
  * Acute myeloid leukemia, acute lymphocytic leukemia, lymphoma, histiocytoses, myelodysplasia, juvenile chronic myelomonocytic leukemia, aplastic anemia, paroxysmal nocturnal hemoglobinuria, or Fanconi's anemia

    * Confirmed by cytochemistry, immunophenotyping, and/or chromosomal abnormalities
  * Multiple myeloma
  * Hereditary immunodeficiency disorders

    * Confirmed by immunologic determination
  * Sickle cell anemia or beta-thalassemia

    * Confirmed by hemoglobin electrophoresis
  * Storage disorders (e.g., Gaucher's disease, Hurler's disease, or metachromatic leukodystrophy)

    * Confirmed by metabolic testing
  * Other non-malignant conditions
* Eligible for allogeneic peripheral blood stem cell or bone marrow transplantation

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing allogeneic blood or marrow stem cell transplantation (alloSCT).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 1996-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Toxicity | 6 months
  Number of irreversible severe (grade 3) or life-threatening or lethal (grade 4-5) organ toxicities.
Time to engraftment | 6 months
  Days from infusion of stem cells to recovery of PMN > 500/ul for two consecutive determinations, transfusion independence for platelets (>20,000/ul) and RBCs (Hct > 25%). The bone marrow function is considered durable if reconstitution persists for at least 6 months.

SECONDARY OUTCOMES:
Clinical response | 6 months
  Number of participants with a partial response (residual though reduced evidence of active disease) and/or complete response (disappearance of all measurable disease, signs, symptoms, and hematologic or biochemical changes related to the disease, for >3 months).
Survival rate | 6 months
Number of participants with Graft-versus-host disease | 6 months
Time to treatment failure and relapse | 6 months
  Time from day 1 of chemoradiotherapy to transplant-related death or disease relapse.

CONTACTS AND LOCATIONS:
Overall Officials: David G. Savage, MD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York, United States